CLINICAL TRIAL: NCT02472977
Title: A Phase 1/2 Study of the Safety and Efficacy of Ulocuplumab Combined With Nivolumab in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Safety and Efficacy Study of Ulocuplumab and Nivolumab in Subjects With Solid Tumors
Acronym: CXCessoR4
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Trial terminated because of lack of efficacy in the short term acute phase
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CA212-115; 2015-000136-15 (EudraCT Number)
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Solid Tumor
MeSH Terms: interventions — ulocuplumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-936564 (Ulocuplumab) + Nivolumab, Tumor type arm (SCLC) (Active Comparator): Small cell lung cancer (SCLC)
  Interventions: Drug: Ulocuplumab; Drug: Nivolumab
- BMS-936564 (Ulocuplumab) + Nivolumab, Tumor type arm (PAC) (Active Comparator): Pancreatic cancer (PAC)
  Interventions: Drug: Ulocuplumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ulocuplumab
  Other Names: BMS-936564
Drug: Nivolumab

SUMMARY:
The purpose of this study is to determine whether the combination of Ulocuplumab and Nivolumab is safe and effective in the treatment of pancreatic cancer and small cell lung cancer.

DETAILED DESCRIPTION:
* Intervention model: Single group for Stage 1 DLT, then Parallel
* Data Monitoring Committee: No (Stage 1) Yes (Stage 2 Randomized Ph2)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* SCLC or PAC that is advanced or has spread to other parts of the body
* Treated with at least one other chemotherapy that did not work or where cancer relapsed
* Minimal limitations on activities of daily living as measured by Eastern Cooperative Oncology Group (ECOG) score of 0-1

Exclusion Criteria:

* Patients with cancer that spread to the brain
* Active, known or suspected autoimmune disease
* Prior treatment with any drug that targets T cell co-stimulation pathways (such as checkpoint inhibitors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (6):
  - University Of Colorado Hosp, Aurora, Colorado
  - Indiana University Health, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Columbia University Medical Center (Cumc), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Local Institution, Helsinki, Finland

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 61 participants were enrolled; 41 participants entered the treatment period.
Groups:
- PAC DL1 (DLT): Pancreatic Adenocarcinoma (PAC) Dose level 1, 400 mg ulocuplumab QW + 3 mg/kg nivolumab Q2W
- PAC DL-1 (Tot): Pancreatic Adenocarcinoma (PAC) Dose level -1, 200 mg ulocuplumab QW + 3 mg/kg nivolumab Q2W
- SCLC (Tot): All Small Cell Lung Cancer (SCLC) subjects in study, 1 subject received 400 mg ulocuplumab QW + 3 mg/kg nivolumab Q2W and 7 subjects received 200 mg ulocuplumab QW + 3 mg/kg nivolumab Q2W
Period: Overall Study
Arm/Group | PAC DL1 (DLT) | PAC DL-1 (Tot) | SCLC (Tot)
Started | 6 | 27 | 8
Completed | 0 | 0 | 0
Not Completed | 6 | 27 | 8
Not completed — Disease progression | 4 | 25 | 6
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Study drug toxicity | 2 | 0 | 2
Not completed — Subject request to discontinue treatment | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | PAC DL1 (DLT) | PAC DL-1 (Tot) | SCLC (Tot) | Total
Number analyzed (Participants) | 6 | 27 | 8 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All treated participants
  years | 63.3 (5.05) | 61.9 (7.93) | 60.1 (14.13) | 61.7 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    Female | 1 | 14 | 4 | 19
    Male | 5 | 13 | 4 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    Hispanic or Latino | 0 | 1 | 1 | 2
    Not Hispanic or Latino | 6 | 22 | 7 | 35
    Unknown or Not Reported | 0 | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 2 | 1 | 3
    White | 6 | 25 | 7 | 38
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and Immune-mediated AEs
Description: The number participants who experienced on-study AEs, SAEs, and AEs requiring immune modulating medication is reported.
Time Frame: From first dose until date of last dose of ulocuplumab or nivolumab plus 100 days (assessed up to January 2017, approximately 18 months)
Population: All treated participants. Participants in the SCLC (Tot) Arm were not evaluated for Immune-mediated AEs
Measure: Number; unit: Participants
Arm/Group | PAC DL1 (DLT) | PAC DL-1 (Tot) | SCLC (Tot)
Number analyzed (Participants) | 6 | 27 | 8
Participants
  Adverse Events | 6 | 27 | 8
  Serious Adverse Events | 3 | 21 | 7
  Immune-mediated AEs: number analyzed (Participants) | 6 | 27 | 0
  Immune-mediated AEs | 1 | 3 |

2. Primary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 Criteria
Description: ORR is defined as the number of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of treated participants. BOR is defined as the best response designation recorded between the first dose date and the date of progression per RECIST 1.1, or the date of subsequent anti-cancer therapy, whichever occurs first. CR= Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD)=At least a 20% increase in the sum of diameters of target lesions, referencing the smallest sum on study, and an absolute increase of at least 5 mm, or the appearance of one or more new lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, referencing the smallest sum diameters while on study.
Time Frame: From first dose until disease progression or treatment discontinuation (assessed up to January 2017, approximately 18 months)
Population: All treated participants in PAC arms. ORR data was not collected for SCLC arm.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | PAC DL1 (DLT) | PAC DL-1 (Tot) | SCLC (Tot)
Number analyzed (Participants) | 6 | 27 | 0
Percentage of participants | 0 [0 to 39.3] | 0 [0 to 10.5] |

3. Primary Outcome: Overall Survival (OS)
Description: If a Phase 2 comparative study is initiated and, for PAC only: Overall Survival is defined as the time from randomization to date of death due to any cause.
Time Frame: From date of randomization to date of death (assessed up to study completion, approximately 18 months)
Population: OS data was not collected for any participants
Arm/Group | PAC DL1 (DLT) | PAC DL-1 (Tot) | SCLC (Tot)
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: The number of participants who experienced on-study Grade 3 or 4 laboratory abnormalities (without Grade 3 or 4 abnormality at baseline) was reported for each arm.
Time Frame: as for outcome 1
Population: All treated participants in PAC arms. Lab abnormality data was not collected for SCLC arm.
Measure: Number; unit: Participants
Arm/Group | PAC DL1 (DLT) | PAC DL-1 (Tot) | SCLC (Tot)
Number analyzed (Participants) | 6 | 27 | 0
Participants
  Increased lymphocytes | 1 | 2 |
  Decreased platelet count | 1 | 2 |
  Hemoglobin | 1 | 1 |
  Leukocytes | 0 | 1 |
  Neutrophils | 0 | 0 |
  Platelet Count | 1 | 2 |
  Alanine Aminotransferase | 0 | 3 |
  Alkaline Phosphatase | 1 | 11 |
  Aspartate Aminotransferase | 0 | 5 |
  Bilirubin | 0 | 1 |
  Creatine | 0 | 0 |
  Hypernatremia | 0 | 0 |
  Hyponatremia | 1 | 3 |
  Hypermagnesemia | 0 | 0 |
  Hypomagnesemia | 0 | 0 |
  Hypercalcemia | 0 | 0 |
  Hypocalcemia | 0 | 0 |
  Hyperkalemia | 0 | 1 |
  Hypokalemia | 0 | 0 |
  Amylase | 1 | 0 |
  Lipase | 1 | 1 |

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival is defined as the time from first dosing date to the date of the first documented tumor progression, as determined by the investigator according to RECIST 1.1 criteria, or death due to any cause, whichever occurs first. Participants who die without a reported prior progression will be considered to have progressed on the date of their death. PFS was not assessed for this study due to the small number of participants.
Time Frame: From first dose to date of progression (assessed up to January 2017, approximately 18 months)
Population: PFS data was not collected for any participants
Arm/Group | PAC DL1 (DLT) | PAC DL-1 (Tot) | SCLC (Tot)
Number analyzed (Participants) | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Electrocardiogram Abnormalities
Description: The number of participants experiencing electrocardiogram abnormalities was reported for each arm
Time Frame: From first dose to date of last dose plus 30 days
Population: Electrocardiogram data was not collected for any participants
Arm/Group | PAC DL1 (DLT) | PAC DL-1 (Tot) | SCLC (Tot)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to date of last dose of ulocuplumab or nivolumab plus 100 days (assessed up to January 2018, approximately 18 months)
Arm/Group | PAC DL1 (DLT) | PAC DL-1 (Tot) | SCLC (Tot)
All-Cause Mortality (participants affected / at risk) | 3/6 | 16/27 | 5/8
Serious Adverse Events (participants affected / at risk) | 3/6 | 21/27 | 7/8
Other Adverse Events (participants affected / at risk) | 6/6 | 26/27 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PAC DL1 (DLT) (N=6) | PAC DL-1 (Tot) (N=27) | SCLC (Tot) (N=8)
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 16 | 3
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 2 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PAC DL1 (DLT) (N=6) | PAC DL-1 (Tot) (N=27) | SCLC (Tot) (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 | 6 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 7 | 1
Tachycardia (Cardiac disorders) | 0 | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 0
Ascites (Gastrointestinal disorders) | 1 | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 5 | 1
Chills (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 11 | 2
Pain (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 5 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 6 | 2
Amylase increased (Investigations) | 2 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 4 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 6 | 0
Blood bilirubin increased (Investigations) | 0 | 3 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 2
C-reactive protein increased (Investigations) | 0 | 2 | 0
Lipase abnormal (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 3
Platelet count decreased (Investigations) | 0 | 4 | 0
Troponin increased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 3 | 1
White blood cell count increased (Investigations) | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-01-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT02472977/SAP_000.pdf
  • Study Protocol (2016-01-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT02472977/Prot_001.pdf